CLINICAL TRIAL: NCT01114438
Title: Post Marketing Study in Subjects Who Have Type 2 Diabetes Using the EndoBarrier™ Gastrointestinal Liner
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Morphic Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-1
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Results first posted 2017-02-20 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device (Experimental)
  Interventions: Device: EndoBarrier Gastrointestinal Liner

INTERVENTIONS:
Device: EndoBarrier Gastrointestinal Liner — EndoBarrier Gastrointestinal Liner is intended to remain in vitro for 12 months.

SUMMARY:
The purpose of this study is to evaluate EndoBarrier Gastrointestinal Liner in the post marketing environment in subjects who are obese and have Type 2 Diabetes.

DETAILED DESCRIPTION:
Patients with obesity are at significantly greater risk of developing complications such as pulmonary dysfunction, diabetes, hypertension, and other co-morbid risks. NIH panel recommendations state that even a 10% short-weight loss would greatly reduce these risks. GI Dynamics' EndoBarrier represents a viable alternative to other short-term pre-surgical weight loss methods. EndoBarrier is a device that can be implanted and removed through minimal invasive endoscopic techniques. This endoscopic procedure brings potential benefits to patients in that it is minimally invasive, efficacious, and allows patients to recover faster with less morbidity and mortality

ELIGIBILITY:
Inclusion Criteria:

* Subjects Age > 18 years and ≤65 years - Male or Female
* Subjects with Type 2 Diabetes > 1 and ≤ 10 years in duration
* Subjects with an Hb A1c level > 7.5 and ≤ 10.0
* Subjects taking oral Type 2 Diabetes medications and/or insulin. Metformin is allowed, but not required.
* Subjects with a BMI > 30 and< 50
* Subjects willing to comply with study requirements
* Subjects who have signed an informed consent form
* Women who are post-menopausal, surgically sterile or on contraceptives and agree to remain on contraceptives for the duration of their study participation and agree not to become pregnant during the study.

Exclusion Criteria:

* Subjects taking Inhibitors of dipeptidyl peptidase 4 inhibitors (ie. Januvia (sitagliptin), Galvus (vildagliptin) or incretins (ie. Byetta (exenatide), Victoza (liraglutide)
* Subjects requiring insulin >150 units per day

  • Subjects with probable insulin production failure (fasting C Peptide serum <1.0 ng/mL)
* Subjects diagnosed with Type 1 Diabetes Mellitus or having a history of ketoacidosis
* Subjects requiring NSAIDs (non-steroidal anti-inflammatory drugs) or prescription anticoagulation therapy during the implant period
* Subjects with or a history of iron deficiency and/or iron deficiency anemia
* Subjects with or a history of abnormalities of the GI tract
* Subjects with symptomatic gallstones or kidney stones at the time of screening
* Subjects with a known infection
* Subjects with or a history of coagulopathy, upper gastro-intestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasia
* Subjects mentally retarded or emotionally unstable, or exhibits psychological characteristics which, in the opinion of the Investigator, makes the subject a poor candidate for device placement or clinical study participation
* Subjects with previous GI surgery that could affect the ability to place the device or the function of the implant
* Subjects with active H. pylori (Note: Subjects may be enrolled if they had a prior history of H. Pylori and were successfully treated. If Subjects have active H. pylori at baseline, they can receive appropriate treatment and then subsequently enroll to the study.)
* Subject or Family history of a known diagnosis or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder
* Subjects with active and uncontrolled gastroesophageal reflux disease (GERD)
* Subjects with severe liver or kidney failure (serum creatinine >180mmol/l)
* Subjects with poor dentition who can not adequately chew their food

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Teare, MD, Principal Investigator — Imperial College/St. Mary's Hospital
Locations (3):
- United Kingdom (3):
  - Imperial College/St. Mary's Hospital, London
  - Trafford General Hospital/NOSC, Manchester
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual subject data is on file at the Sponsor

RESULTS

PARTICIPANT FLOW:
Groups:
- EndoBarrier Gastrointestinal Liner: EndoBarrier Gastrointestinal Liner: EndoBarrier Gastrointestinal Liner is intended to remain in vitro for 6 months.
Period: Overall Study
Arm/Group | EndoBarrier Gastrointestinal Liner
Started | 45
Completed | 31
Not Completed | 14
Not completed — Adverse Event | 10
Not completed — concomitant medication | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | EndoBarrier Gastrointestinal Liner
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (7.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 45
Region of Enrollment [Number; unit: participants]
  United Kingdom | 45
Weight (kg) [Mean (Standard Deviation); unit: kg] | 115 (21.02)
BMI [Mean (Standard Deviation); unit: kg/m2] | 40.0 (5.79)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 4.6 (2.79)
Baseline HbA1c [Mean (Standard Deviation); unit: %] | 8.5 (0.85)
Baseline glucose [Mean (Standard Deviation); unit: mmol/L] | 9.5 (2.95)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c (%) Measured at Week 52
Time Frame: 12 months
Population: Analysis was conducted on the Full Analysis Set (FAS) defined as all subjects enrolled and implanted with the EndoBarrier, There were 29 subjects' data available for analysis of HbA1c at the defined 12 month (week 52) endpoint.
Measure: Median (Full Range); unit: % glycated hemoglobin
Groups:
- EndoBarrier Liner Device: EndoBarrier Gastrointestinal Liner: EndoBarrier Gastrointestinal Liner is intended to remain in vitro for 6 months.
Arm/Group | EndoBarrier Liner Device
Number analyzed (Participants) | 29
% glycated hemoglobin | 7.3 [5.8 to 11.5]

2. Primary Outcome: Total Weight Change From Baseline to Week 52
Description: Total weight change at 12 months (kg) compared to baseline
Time Frame: 12 months
Population: Analysis was conducted on the Full Analysis Set (FAS) defined as all subjects enrolled and implanted with the EndoBarrier, There were 29 subjects' data available for weight loss analysis at the defined 12 month endpoint.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | EndoBarrier Liner Device
Number analyzed (Participants) | 29
kg | -12.1 (7.0)

3. Primary Outcome: Changes in Diabetic Medications at Treatment Completion Compared to Baseline
Description: number of patients with a decrease, increase or no change in diabetic medications at time of EndoBarrier explantation (treatment completion)
Time Frame: 12 months
Population: Analysis was conducted on subjects with a device
Measure: Count of Participants; unit: Participants
Groups:
- Decrease in Glucose-Lowering Meds: Subjects implanted with device for 12 Months with an Decrease in medication at the time of device removal compared to Baseline medication levels
- Increase in Glucose-Lowering Meds at Week 52: Subjects implanted with device for 12 Months with an Increase in medication at the time of device removal compared to Baseline medication levels
- No Change in Glucose-Lowering Meds at Week 52: Subjects implanted with device for 12 Months with no change in medication at the time of device removal compared to Baseline medication levels
Arm/Group | Decrease in Glucose-Lowering Meds | Increase in Glucose-Lowering Meds at Week 52 | No Change in Glucose-Lowering Meds at Week 52
Number analyzed (Participants) | 45 | 45 | 45
Participants | 23 | 4 | 18

4. Primary Outcome: Change From Baseline in SF 36v2 Quality of Life Assessment
Description: Quality of life was measured using Survey Form SF-36v2 licensed from Quality Metric, Inc (Lincoln, RI). Physical and Mental component scores were measured at baseline, month 12 (at the time of explant) and 6 months post explant with results self-recorded by each subject. The SF-36 v2 physical component summary (PCS) score as well as the mental component summary score (MCS) ranged between 0 and 100, with higher scores reflecting better quality of life in each case.
Time Frame: Baseline, 12 months (explant), 6 months post explant (18 months post baseline)
Population: The number of participants analyzed reflects all participants who received the implant and were assessed for QoL at the respective time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Device at Month 12 (Explant); Device at 6 Months Post-explant: EndoBarrier Gastrointestinal Liner: EndoBarrier Gastrointestinal Liner was implanted in participants for 12 months and then removed
Arm/Group | Device at Month 12 (Explant) | Device at 6 Months Post-explant
Number analyzed (Participants) | 35 | 25
units on a scale
  PCS-Change from Baseline | 1.0 (9.49) | 1.0 (8.33)
  MCS-Change from Baseline | 3.0 (9.66) | -0.5 (14.12)

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Device: EndoBarrier Gastrointestinal Liner: EndoBarrier Gastrointestinal Liner is intended to remain in vitro for 6 months.
Arm/Group | Device
Serious Adverse Events (participants affected / at risk) | 13/45
Other Adverse Events (participants affected / at risk) | 40/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device (N=45)
Atrial Flutter (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Gastrointestinal hemorrhage (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device (N=45)
Anaemia (Blood and lymphatic system disorders) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 18 (22)
Diarrhea (Gastrointestinal disorders) | 9 (10)
Nausea (Gastrointestinal disorders) | 8 (8)
Vomiting (Gastrointestinal disorders) | 8 (10)
Abdominal discomfort (Gastrointestinal disorders) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 5 (5)
Abdominal pain lower (Gastrointestinal disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 4 (4)
Chest pain (General disorders) | 3 (3)
Edema peripheral (General disorders) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 3 (3)
Procedural nausea (Injury, poisoning and procedural complications) | 8 (8)
Procedural vomiting (Injury, poisoning and procedural complications) | 4 (4)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 14 (15)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Depression (Psychiatric disorders) | 5 (5)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less